CLINICAL TRIAL: NCT02798627
Title: A Phase II, Double-Blind, Placebo-Controlled, Trial Of NS2359 For The Treatment of Cocaine Dependence
Brief Title: Trial Of NS2359 For The Treatment of Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Saniona (Industry); The Dana Foundation (Other)
Responsible Party: Principal Investigator, Kyle Kampman, Professor of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 824109
Record Dates: First submitted 2016-05-17; First posted 2016-06-14 (Estimated); Results first posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — GSK372475

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NS2359 (Experimental): The initial dose of the NS2359 will be two mg once daily. Patients with difficult adverse events at the 2 mg dose will be allowed to reduce to 1 mg once daily. Subjects will participate in weekly cognitive behavioral relapse prevention psychotherapy from week 2 through week 9.
  Interventions: Drug: NS2359
- placebo (Placebo Comparator): Placebo pills matched to NS2359 pills will be given once daily. Patients with difficult adverse events at the 2 mg placebo will be allowed to reduce to 1 mg placebo once daily. Subjects will participate in weekly cognitive behavioral relapse prevention psychotherapy from week 2 through week 9.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NS2359 — NS2359 is a small molecule which inhibits the reuptake of dopamine, norepinephrine and serotonin with equal affinity.
  Arms: NS2359
Drug: placebo — Placebo pills identical in appearance to the NS2359 will be provided
  Arms: placebo

SUMMARY:
NS2359 attenuates the euphoria associated with cocaine use. In a manner parallel to cocaine, NS2359 blocks the reuptake of dopamine (DA), norepinephrine (NE), and serotonin (5HT) with nanomolar affinities at the 3 transporters. In primates NS2359 significantly attenuated cocaine self-administration. In several phase II clinical trials for major depressive disorder and adult attention deficit disorder, NS2359 did not cause euphoria. NS2359 exhibited no abuse potential in a human laboratory study comparing NS2359 with amphetamine. In a phase I human laboratory interaction study, NS2359 showed no toxicity after 20 or 40 mg of cocaine, but it attenuated the both the rewarding and cardiovascular effects of intravenous cocaine. On the basis of these promising studies, investigators propose a Phase II double-blind clinical trial of NS2359 in cocaine addiction (CA). The proposed trial will involve 100 CA subjects participating in an eight week trial, including a 1-week baseline and 8 weeks of NS2359 or placebo treatment. Four weeks after completing the medication phase, there will be one follow-up visit. Subjects will be randomly assigned to treatment with placebo or 2 mg NS2359 daily, with a possible decrease to 1 mg daily for adverse events. This dose range is selected on the basis of phase I and II evidence of tolerability and NS2359 plasma levels which were associated with blockade of cocaine reward. This project has the potential to identify the first effective pharmacotherapy for CA.

DETAILED DESCRIPTION:
In this phase II randomized double-blind, placebo-controlled trial, 40 persons will be randomized to NS2359 and 40 to placebo. The primary hypothesis is: more NS2359-treated subjects (compared to placebo-treated subjects) will achieve 3 consecutive weeks of cocaine abstinence, as measured by urine benzoylecgonine (BE) assay, during the last three weeks of the trial. The study is 9 weeks: one week of screening, followed by an 8-week double-blind, placebo-controlled trial. All subjects will receive weekly cognitive behavioral therapy (CBT) to encourage abstinence during their 3 times weekly clinic visits. Investigators expect ~ 20% dropout rate, based on our recent CA clinical trials (eg, Kampman et al, 2015 and 2013), so 80 randomized patients will yield ~ 64 study completers. There will be a 1 month start-up period, followed by 20 months of recruitment for the study. The 1 month start-up period will allow for training of staff, preparation of study capsules, placement of study advertisements, etc. Penn IRB approval has been obtained. There will be a 2-month termination period to allow the final patients to complete the study. Data cleaning, statistical analyses and preparation of reports will be done in the final two months. Based on recent cocaine pharmacotherapy trials conducted by our team, monthly enrollment of ~4 CA participants (respondents to flyers and advertisements) is feasible.

Recruitment will occur at the University of Pennsylvania's Treatment Research Center (TRC), led by Kyle Kampman, MD, and Wade Berrettini, MD, PhD, Professors of Psychiatry at Penn. At the TRC, CA patients are respondents to advertisements for free treatment of CA. The ethnicity is 90% African-American, 9 % European-American, 70% male, mean age 47 (+/- 12).

ELIGIBILITY:
Inclusion Criteria:

1. Male and females, 18-65 years old.
2. Meets diagnostic criteria (DSM-V) for current diagnosis of cocaine use disorder, moderate to severe, by semi-structured interview.
3. In the past 30 days, used no less than $100-worth of cocaine
4. Speaks, understands, and prints in English.

Exclusion Criteria:

1. Meets DSM-V criteria for substance use disorder, moderate to severe, for a substance other than cocaine, alcohol or nicotine. Subjects with comorbid alcohol use disorder will be accepted if their alcohol use disorder is not severe enough to require a medical alcohol detoxification.
2. Needs treatment with any psychoactive medications (with the exception of diphenhydramine or melatonin, if necessary, for sleep).
3. Meets current or lifetime DSM-V criteria for schizophrenia or any psychotic disorder, or organic mental disorder.
4. Has another Axis I psychiatric disorder that in the opinion of the physician will interfere with completion of the study or place the patient at heightened risk through participation in the trial.
5. Has evidence of a history of significant hematological, pulmonary, endocrine, cardiovascular, renal or gastrointestinal disease.
6. Use of an investigational medication in the 30 days prior to randomization.
7. Is female and has a positive pregnancy test, is contemplating pregnancy in the next 6 months, is nursing, or is not using effective contraception (if relevant).

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-05; Primary Completion 2020-03 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wade Berrettini, MD, PhD, Principal Investigator — University of Pennsylvania Perelman School of Medicine, Department of Psychiatry
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment by advertising in local newspapers and radio began in 07/2016 and ended in 12/2018.
Pre-assignment Details: Participants had a screening telephone appointment to determine eligibility. If eligible, they were seen at the clinic for history, physical exam and urine drug screen. A positive urine drug screen for a cocaine metabolite (BE) was used as a stratifying variable in randomization.
Period: Overall Study
Arm/Group | NS2359 | Placebo
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NS2359 | Placebo | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56.4 [49.5 to 59.6] | 52 [49.8 to 56.9] | 53.8 [49.6 to 58.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 24 | 23 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 26 | 50
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55
Days of cocaine use in past 30 [Median (Inter-Quartile Range); unit: Days] | 9.0 [4.0 to 20] | 9.5 [5.0 to 17.0] | 9.0 [5.0 to 17.0]

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Achieved Abstinence From Cocaine During the Last Three Weeks of the Trial
Description: Number of Participants Who Report no Cocaine Use and Have no Cocaine Positive Urine Drug Screens in the NS2359 Group Versus the Placebo Group Comparator During the Last Three Weeks of the Trial [ Time Frame: weeks 6,7.8 of the trial ] Number of subjects with cocaine abstinence as measured through three-times-weekly urine benzoylecgonine (BE) levels in urine drug screen (UDS) and self-reports of use from the Time Line Follow Back. UDS results and TLFB reports combined to yield weekly use/no-use indicators for each week of treatment.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | NS2359 | Placebo
Number analyzed (Participants) | 27 | 28
participants | 2 | 2
Statistical Analysis 1: Comparison: NS2359 vs Placebo; Test type: Superiority; p = 0.97, Chi-squared

2. Secondary Outcome: Average Weekly Cocaine Craving Scores NS2359 Group Versus the Placebo Group Comparator [ Time Frame: Once Per Week in Weeks 2 Through 8 ]
Description: As measured by average weekly scores for cocaine craving on the brief substance craving scale combining cocaine craving frequency, intensity and duration. Minimum value 0 maximum value 12 higher scores indicate worse craving.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | NS2359 | Placebo
Number analyzed (Participants) | 27 | 28
score on a scale | 4.09 (0.39) | 3.89 (0.33)

ADVERSE EVENTS:
Time Frame: Adverse event data was measured over 12 weeks
Description: Patients completed adverse event forms and answered specific questions about adverse events
Arm/Group | NS2359 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 11/27 | 1/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NS2359 (N=27) | Placebo (N=28)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0) — heart racing
flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
sedation (Nervous system disorders) | 3 (3) | 0 (0)
increased blood pressure (Vascular disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Small numbers of individuals analyzed. Some noncompliance per plasma NS2359 levels at mid and end treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT02798627/Prot_SAP_000.pdf